CLINICAL TRIAL: NCT00326027
Title: Profi-Study: Symptom Reduction in Hospitalized Patients Suffering From Symptomatic Non-erosive or Erosive Gastroesophageal Reflux Disease Treated With Pantoprazole 20 or 40 mg o.d. for 7 Days
Brief Title: Efficacy of Pantoprazole in Patients Older Than 18 Years Who Have Symptoms of Non-erosive Reflux or Gastroesophageal Reflux Disease (BY1023/DE-004)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nycomed (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BY1023/DE-004
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Gastroesophageal Reflux
Keywords: GERD; Pantoprazole; NERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pantoprazole 20 mg
  Interventions: Drug: Pantoprazole
- 2 (Active Comparator): Pantoprazole 40 mg
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Efficacy of Pantoprazole

SUMMARY:
The aim of the study is to evaluate the effect of pantoprazole on fast symptom reduction in hospitalized patients with NERD (non-erosive reflux disease) or GERD (gastroesophageal reflux disease, Los Angeles [LA] Grade A-D). During the study, the patients will complete a patient-orientated, self-assessed reflux questionnaire (ReQuest™). The study duration consists of a treatment period of 7 days ± 3 days. Pantoprazole (tablet) will be administered once daily in the morning to patients with NERD or GERD at one dose level for each indication. The study will provide further data on the safety and tolerability of pantoprazole.

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent
* Inpatients (hospitalization during the entire study period is mandatory)
* Symptomatic (heartburn, acid regurgitation or dysphagia for at least 1 day since admission to the hospital) non-erosive reflux disease (NERD) or erosive gastroesophageal reflux disease (GERD, LA Grade A-D)

Main Exclusion Criteria:

* Known Zollinger-Ellison syndrome or other gastric hypersecretory condition
* Previous acid-lowering surgery or other surgery of the esophagus and/or upper gastrointestinal tract (exception: polypectomy and cholecystectomy)
* On initial endoscopy, presence of obstructive esophageal strictures, Schatzki's ring, esophageal diverticula, esophageal varices, achalasia or Barrett's esophagus with known high-grade dysplasia or longer than 3 cm
* Acute peptic ulcer and/or ulcer complications
* Pyloric stenosis
* Known inflammatory bowel diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Symptom reduction from reflux disease related symptoms as measured by the questionnaire ReQuest™-GI (gastrointestinal) after 1 day of treatment | 1 day

SECONDARY OUTCOMES:
Symptom reduction from reflux disease related symptoms as measured by the questionnaire ReQuest™-GI (gastrointestinal) after 2 to 7 days of treatment | 7 days
Symptom relief rates as measured by ReQuest™ after 7 days of treatment | 7 days
Safety | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Mössner, Prof., Principal Investigator — Universitätsklinikum Leipzig, Leipzig, Germany
Locations (32):
- Germany (32):
  - Nycomed Deutschland GmbH, Augsburg
  - Nycomed Deutschland GmbH, Berlin
  - Nycomed Deutschland GmbH, Brandenburg
  - Nycomed Deutschland GmbH, Cologne
  - Nycomed Deutschland GmbH, Erlangen
  - Nycomed Deutschland GmbH, Frankfurt
  - Nycomed Deutschland GmbH, Gera
  - Nycomed Deutschland GmbH, Göttingen
  - Nycomed Deutschland GmbH, Greifswald
  - Nycomed Deutschland GmbH, Halle
  - Nycomed Deutschland GmbH, Hamburg
  - Nycomed Deutschland GmbH, Ingolstadt
  - Nycomed Deutschland GmbH, Jena
  - Nycomed Deutschland GmbH, Kassel
  - Nycomed Deutschland GmbH, Kiel
  - Nycomed Deutschland GmbH, Leipzig
  - Nycomed Deutschland GmbH, Ludwigsburg
  - Nycomed Deutschland GmbH, Ludwigshafen
  - Nycomed Deutschland GmbH, Lübeck
  - Nycomed Deutschland GmbH, Mainz
  - Nycomed Deutschland GmbH, Marburg
  - Nycomed Deutschland GmbH, Minden
  - Nycomed Deutschland GmbH, München
  - Nycomed Deutschland GmbH, Münster
  - Nycomed Deutschland GmbH, Neubrandenburg
  - Nycomed Deutschland GmbH, Offenbach
  - Nycomed Deutschland GmbH, Oldenburg
  - Nycomed Deutschland GmbH, Recklinghausen
  - Nycomed Deutschland GmbH, Rostock
  - Nycomed Deutschland GmbH, Stade
  - Nycomed Deutschland GmbH, Weimar
  - Nycomed Deutschland GmbH, Wiesbaden